CLINICAL TRIAL: NCT01848691
Title: Phase 1 Study of Carbon Monoxide Monitor for the Measurement of End-Tidal Carbon Monoxide Levels in Children With or Without Hemolysis
Brief Title: Carbon Monoxide Monitor for the Measurement of End-Tidal Carbon Monoxide Levels in Children With or Without Hemolysis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ashutosh Lal (Other)
Responsible Party: Sponsor-Investigator, Ashutosh Lal, Associate Hematologist/Oncologist, UCSF Benioff Children's Hospital Oakland
Organization: UCSF Benioff Children's Hospital Oakland (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: Capnia CoSense Award 12.8062
Record Dates: First submitted 2013-05-03; First posted 2013-05-07 (Estimated); Last update posted 2014-06-02 (Estimated); Status verified 2014-05

CONDITIONS: Sickle Cell Anemia
MeSH Terms: conditions — Anemia, Sickle Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sickle Cell (Experimental): This arm will include 20 children with sickle cell anemia
  Interventions: Other: Measurement of carbon monoxide level in exhaled breath
- Control (Active Comparator): This arm will include 20 children without sickle cell anemia
  Interventions: Other: Measurement of carbon monoxide level in exhaled breath

INTERVENTIONS:
Other: Measurement of carbon monoxide level in exhaled breath — Measurement of end-tidal carbon monoxide concentration
  Other Names: CoSense Carbon Monoxide Monitor

SUMMARY:
People who have Sickle Cell Anemia (HbSS) produce red blood cells with shorter lifespans. These red blood cells breakdown faster, and this is called hemolysis. When red blood cells breakdown, a tiny amount of Carbon Monoxide (CO) is released into the blood and is eliminated in exhaled breath. This research study will use a device called CoSense™, which will measure Carbon Monoxide (CO) levels in breath. The purpose of the study is to see how well the device measures the CO levels that an individual breathes out.

DETAILED DESCRIPTION:
Subjects diagnosed with homozygous sickle cell anemia (Hb SS) have red blood cells with a decreased lifespan, which leads to an increase in the rate of heme turnover. Carbon monoxide (CO) is a by-product of heme oxidation and is excreted in exhaled breath. The concentration of CO in end-tidal breath can be measured and used to indicate the rate of heme oxidation, bilirubin production and the presence of hemolysis. The objective of this study is to characterize the performance of CoSense™ in children with or without sickle cell anemia. This is a single-center, open-label, non-randomized, proof of concept study to characterize the ability of CoSense™ to assess ETCO levels in subjects with a diagnosis of sickle cell anemia (Hb SS). Up to 40 children (5-14 years old), of which 20 participants will have a diagnosis of Hb SS, will be enrolled. Each participant will have two breath samples collected non-invasively, one immediately after the other. It takes approximately 120 seconds to collect the each breath sample. This study and investigational device are a non-significant risk to the patient. The nasal cannula is made of a biocompatibility-tested polyvinyl chloride (PVC) material with a soft open-end, and will be gently placed adjacent to one of the nostrils and partially inserted by approximately 5 mm. The objective of this study will be assessed through reproducibility of ETCO measurements and comparison of ETCO levels between children diagnosed with Hb SS and healthy children. The study would help in the development of a portable CO measurement device which has potential health applications in monitoring diseases with altered bilirubin metabolism.

ELIGIBILITY:
Inclusion Criteria:

* Parental / legal guardian consent
* Subject assent for participants ages 7 and above
* Male and female children ages 5 - 14 years old
* For Hb SS subjects, hemoglobin ≤ 10 g/dL (based on a laboratory tests performed over the last 6 months and confirmed within 4 weeks prior to breath collection, as part of the subject's clinical care)

Exclusion Criteria:

* For healthy subjects, known to have the sickle cell trait
* Had a red blood cell transfusion within 12 weeks prior to enrollment
* Currently a primary smoker or was a primary smoker within 4 weeks prior to enrollment
* Exposed to second hand smoke within 24 hours prior to breath sample collections
* Have an upper respiratory infection within 2 weeks of ETCO measurements

Ages: 5 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2012-10; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
End-Tidal Carbon Monoxide Concentration | one year

CONTACTS AND LOCATIONS:
Overall Officials: Ashutosh Lal, MD, Principal Investigator — Children's Hospital & Research Center at Oakland
Locations (1):
- Children's Hospital & Research Center Oakland, Oakland, California, United States